CLINICAL TRIAL: NCT03099837
Title: Maternal and Infant Health Survey
Brief Title: Tongji Maternal and Child Health Cohort
Acronym: TMCHC
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Huazhong University of Science and Technology (Other)
Collaborators: Maternal and Child Health Hospital of Hubei Province (Other); Wuhan Central Hospital (Other); Wuhan Maternal and Child Health Hospital (Unknown)
Responsible Party: Principal Investigator, Nianhong Yang, Professor, Huazhong University of Science and Technology
Other Study IDs: HuazhongU-2013-02
Record Dates: First submitted 2017-03-17; First posted 2017-04-04 (Actual); Last update posted 2020-08-04 (Actual); Status verified 2020-08

CONDITIONS: Weight Gain; Maternal; Diabetes Mellitus, Affecting Fetus; Diet Habit; Pregnancy Complications; Birth Outcomes; Breast Feeding; Growth and Development
MeSH Terms: conditions — Weight Gain; Diabetes Mellitus; Feeding Behavior; Pregnancy Complications; Breast Feeding

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Pregnant mothers
- infants
- children

SUMMARY:
This is a population-based study to obtain data for the evaluation of current used recommendations for weight gain during pregnancy released by IOM (2007) and investigate the association between maternal diet and the health outcomes of mother and offspring.

DETAILED DESCRIPTION:
This is an ongoing population-based prospective cohort study to obtain data for the evaluation of current used recommendations for weight gain during pregnancy released by IOM (2007) and investigate the association between maternal diet and the health outcomes of mother and offspring. 8649 pregnant have been recuited from the first trimester of pregnancy. All datas including the general information, sociodemographic facts, physical exam (body weight, height, blood pressure, etc), laboratory test (hemoglobin, glucose concentration, etc.) and dietary survey (FFQ, 24h food recall) have been collected during the cohort study. Blood sample leftover from the clinical use are remained and stored at -80℃for further measurements. Obstetric characteristics, maternal and perinatal outcomes have been observed and recorded. Growth and development paremeters such as weight, length and head circumference as well as disease information of infants have been collected , feeding pattern and feeding history will be surveyed. All data collected will be used for group analysis only and all private and individual records will be kept secret.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women attending the first visit (<16 weeks ) at at a maternity clinic in one of these following hospitals in Wuhan, China: HMCHH, CHW,WMCHH,JMCHH.

Intention to visit the maternity clinic regularly in HMCHH or CHW or WMCHH or JMCHH.

* Intention to eventually deliver in HMCHH or CHW or WMCHH.
* The pregnant woman and her husband are Chinese.

Exclusion Criteria:

* Pregnant women on chemotherapy.
* Exclude women on certain medications - e.g. psychotropic drugs.
* Exclude women with significant medical conditions e.g. psychosis etc.

Sex: Female
Age Groups: Child, Adult, Older Adult
Study Population: The Tongji Maternal and Child Health enrolled healthy pregnant women at 8-16 weeks gestation when they attended their first antenatal visit at a maternity clinic in one of these following hospitals in Wuhan, China: Hubei Maternal and Child Health Hospital (HMCHH), The Central Hospital of Wuhan(CHW), Wuhan Maternal and Child Health Hospital (WMCHH), Jiang'an Maternal and Child Health Hospital(JMCHH). Babies born from these mothers will be followed up until the child is at least 10 years of age.
Sampling Method: Probability Sample
Enrollment: 8649 (Actual)
Dates: Start 2013-01-10 (Actual); Primary Completion 2023-01-10 (Estimated); Study Completion 2023-01-10 (Estimated)

PRIMARY OUTCOMES:
Effect of weight gain during pregnancy on maternal and child health | During pregnancy, infancy period and childhood, assessed up to 120 months
  To regularly measure the weight gains of pregnant women during pregnancy, and examine their association with maternal and child health.
Effect of factors in pregnancy and early postpartum period on maternal health | During pregnancy and postpartum period, assessed up to 12 months
  To examine the role of maternal nutrition, lifestyle, emotional health, and other environmental factors in pregnancy or postpartum period that can influence future maternal risk of metabolic disorders and even lead to complications of pregnancy, such as gestational diabetes mellitus.
Influence of prenatal and early postnatal factors on child health | During pregnancy, infancy period and childhood, assessed up to 120 months
  To examine the role of maternal nutrition, lifestyle, emotional health, breastfeeding, and other environmental factors in infancy that can influence the development of phenotypes in childhood which confer risk for later metabolic and mental disorders.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kong M, Zhong C, Gao Q, Zhou X, Chen R, Xiong G, Hao L, Yang X, Lu Z, Yang N. Association of elevated mid-pregnancy maternal plasma ferritin concentrations and triglyceride concentrations with the risk of gestational diabetes mellitus: A prospective cohort study. Diabetes Metab Res Rev. 2023 Sep;39(6):e3637. doi: 10.1002/dmrr.3637. Epub 2023 Apr 13. PMID 36958940
- [Derived] Zhong C, Xiong G, Lin L, Li Q, Chen X, Zhang X, Zhang Y, Xu S, Wang X, Gao D, Wu M, Yang S, Han W, Sun G, Yang X, Hao L, Jin Z, Yang N. The association of maternal vaginal bleeding and progesterone supplementation in early pregnancy with offspring outcomes: a prospective cohort study. BMC Pregnancy Childbirth. 2022 May 5;22(1):390. doi: 10.1186/s12884-022-04711-1. PMID 35513779
- [Derived] Li Y, Zhou X, Zhang Y, Zhong C, Huang L, Chen X, Chen R, Wu J, Li Q, Sun G, Yin H, Xiong G, Hao L, Yang N, Yang X. Association of Maternal Dietary Patterns With Birth Weight and the Mediation of Gestational Weight Gain: A Prospective Birth Cohort. Front Nutr. 2021 Nov 26;8:782011. doi: 10.3389/fnut.2021.782011. eCollection 2021. PMID 34901129
- [Derived] Xiong T, Wu Y, Huang L, Chen X, Zhang Y, Zhong C, Gao Q, Hong M, Hu X, Yang X, Yang N, Hao L. Association of the maternal serum albumin level with fetal growth and fetal growth restriction in term-born singletons: a prospective cohort study. Fertil Steril. 2022 Feb;117(2):368-375. doi: 10.1016/j.fertnstert.2021.09.016. Epub 2021 Oct 20. PMID 34686372
- [Derived] Gao Q, Zhong C, Zhou X, Chen R, Xiong T, Hong M, Li Q, Kong M, Xiong G, Han W, Sun G, Yang X, Yang N, Hao L. Inverse association of total polyphenols and flavonoids intake and the intake from fruits with the risk of gestational diabetes mellitus: A prospective cohort study. Clin Nutr. 2021 Feb;40(2):550-559. doi: 10.1016/j.clnu.2020.05.053. Epub 2020 Jun 13. PMID 32593522
- [Derived] Zhou X, Chen R, Zhong C, Wu J, Li X, Li Q, Cui W, Yi N, Xiao M, Yin H, Xiong G, Han W, Hao L, Yang X, Yang N. Fresh fruit intake in pregnancy and association with gestational diabetes mellitus: A prospective cohort study. Nutrition. 2019 Apr;60:129-135. doi: 10.1016/j.nut.2018.09.022. Epub 2018 Oct 24. PMID 30572275